CLINICAL TRIAL: NCT00905060
Title: PHASE 2, Multi-center, Single Arm Investigation of HSPPC-96 Vaccine With Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: HSPPC-96 Vaccine With Temozolomide in Patients With Newly Diagnosed GBM
Acronym: HeatShock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Principal Investigator, Orin Bloch, MD, Principal Investigator, University of California, San Francisco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 081010; C-100-37 (Other: Agenus); NCI-2015-01229 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); NCT00912951 (obsolete NCT alias)
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: Newly Diagnosed Glioblastoma Multiforme, vaccine
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — vitespin; Heat-Shock Response; Temozolomide; Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Protein Peptide-Complex (HSPPC-96) (Experimental): Patients will receive 4 weekly injections of HSPPC-96 followed by a 5th vaccine injection on the same day of the start of maintenance temozolomide administered 2 weeks (+ 4 days) following vaccine administration #4 on the same day of the start of maintenance temozolomide (Day 36). Monthly vaccine injections will then begin on day 21 (+/- 7 days) of the first 28 day temozolomide cycle (Day 56 of the study), 3 weeks following vaccine administration #5 and will continue every 28 days until depletion of vaccine or progression.
  Interventions: Biological: HSPPC-96; Drug: Temozolomide; Procedure: Standard Surgical Resection

INTERVENTIONS:
Biological: HSPPC-96 — Autologous tumor-derived heat shock protein peptide-complex (HSPPC-96) administered at 25 μg per dose injected intradermally once weekly for 4 consecutive weeks and monthly following standard treatment with radiation and temozolomide.
  Other Names: Heat Shock; Vitespen
Drug: Temozolomide — Maintenance temozolomide treatment is given 2 weeks after administration of the fourth vaccine at an initial dose of 150 mg per square meter (mg/m2) for 5 consecutive days in a 28-day cycle. The dose was increased to 200 mg/m2 for 5 days in subsequent cycles.
  Other Names: Temodar
Procedure: Standard Surgical Resection — Patients will undergo standard surgical resection of intracranial tumor
  Other Names: Craniotomy

SUMMARY:
This phase II trial studies the side effects and how well HSPPC-96 (vitespen) and temozolomide work in treating patients with newly diagnosed glioblastoma multiforme. Vaccines made from a person's tumor cells and heat shock protein peptide may help the body to build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving HSPPC-96 (vitespen) together with temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety profile of HSPPC-96 (vitespen) administered concurrently with temozolomide in patients with newly diagnosed glioblastoma multiforme (GBM).

II. To evaluate survival in patients treated with an autologous tumor-derived heat shock protein peptide-complex (HSPPC-96) with concurrent temozolomide.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival (PFS) from date of surgical resection. II. To evaluate the immunologic response to vaccine treatment in a subset of evaluable patients.

OUTLINE:

Approximately 2-5 weeks after standard radiation therapy and temozolomide completion, patients receive vitespen intradermally (ID) on days 1, 8, 15, and 22. Beginning 2 weeks after the 4th dose of vitespen, patients receive a 5th dose of vitespen ID and maintenance temozolomide orally (PO) on days 1-5 (of 28 day courses). On day 21 of course 1, patients receive the 6th dose of vitespen ID and continue vaccinations monthly. Courses repeat every 28 days in the absence of vaccine depletion, disease progression, or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Pre-surgery tissue acquisition Inclusion criteria

1. Age > or equal to 18 years old
2. Life expectancy of greater than 12 weeks.
3. Able to read and understand the informed consent document; must sign the informed consent
4. Must have suspected diagnosis of Glioblastoma Multiforme with a surgical intent to resect at least 90% of enhancing disease
5. Must be eligible for post-surgical treatment with radiotherapy and temozolomide

Post-radiation therapy/pre-vaccine eligibility Inclusion criteria

1. Agree to use contraception or abstain from sexual activity from the time of consent through 1 month after the end of study drug administration
2. Negative serum pregnancy test for female patients of childbearing potential
3. Patients with histologically proven, non-progressive glioblastoma multiforme (GBM)
4. Patient must have received standard of care radiation and temozolomide therapy
5. Must have undergone a at least a 90% resection (determined by the principal investigator (PI)) measured by postoperative magnetic resonance imaging (MRI) scan, T1-weighted contrast scan, or CT scan if clinically indicated, performed within 72 hours after surgery
6. All radiotherapy must be discontinued at least 2 weeks and no more than 5 weeks prior to the first planned vaccine administration
7. Availability of at least 4 doses of vaccine (at least 4 vials for clinical administration produced from the tumor provided)
8. Karnofsky functional status rating > or equal to 70
9. Adequate bone marrow function including the absence of lymphopenia (ANC > 1,500/ mm3; absolute lymphocyte count (ALC) > 500/mm3 ; platelet count >100,000/mm3), adequate liver function (serum glutamic oxaloacetic transaminase/ aspartate aminotransferase (AST), alanine amino transferase (ALT), and alkaline phosphatase <2.5 times institutional upper limit of normals [IULNs] and bilirubin (total) <1.5 mg*IULN), and adequate renal function (BUN and creatinine <1.5 times IULNs

Exclusion Criteria:

Pre-surgery tissue acquisition

1. Current diagnosis of Human Immunodeficiency Virus (HIV testing is not required per protocol)
2. Any prior diagnosis of any other cancer or other concurrent malignancy, with the exception of adequately treated nonmetastatic in situ carcinoma of the uterine cervix or nonmetastatic nonmelanoma skin cancer unless in complete remission and off all therapy for that disease for a minimum of 5 years
3. Any systemic autoimmune disease (e.g., Hashimoto's thyroiditis) and/or any history of primary or secondary immunodeficiency
4. Any prior therapy for glioma
5. Planned use or current use of other investigational therapy for the treatment of glioma

Post-radiation therapy/pre-vaccine Exclusion

1. Inability to comply with study-related procedures
2. Prior diagnosis of any other cancer or other concurrent malignancy, with the exception of adequately treated nonmetastatic in situ carcinoma of the uterine cervix or nonmetastatic nonmelanoma skin cancer unless in complete remission and off all therapy for that disease for a minimum of 5 years
3. Current or active use of chemotherapy (except temozolomide) or immune therapy
4. Contrast MRI findings (or CT scan if MRI is clinically contraindicated) consistent with progression per protocol defined modified Response assessment in neuro-oncology criteria (RANO) criteria. Progression prior to vaccination as determined by the Principal Investigator
5. Patients with active uncontrolled infection
6. Evidence of bleeding diathesis
7. Unstable or severe intercurrent medical conditions
8. Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06-29 (Actual); Primary Completion 2014-06-03 (Actual); Study Completion 2014-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, Principal Investigator — University of California, San Francisco
Locations (9):
- United States (9):
  - University of California, San Francisco, San Francisco, California
  - University of Miami, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Valley Hospital, Paramus, New Jersey
  - Northern Westchester Hospital, Mount Kisco, New York
  - Columbia University, New York, New York
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bloch O, Lim M, Sughrue ME, Komotar RJ, Abrahams JM, O'Rourke DM, D'Ambrosio A, Bruce JN, Parsa AT. Autologous Heat Shock Protein Peptide Vaccination for Newly Diagnosed Glioblastoma: Impact of Peripheral PD-L1 Expression on Response to Therapy. Clin Cancer Res. 2017 Jul 15;23(14):3575-3584. doi: 10.1158/1078-0432.CCR-16-1369. Epub 2017 Feb 13. PMID 28193626

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place between June 29, 2009 and April 2012 for participants scheduled for gross total resection of recurrent Glioblastoma multiforme (GBM) across 8 sites
Period: Surgical Resection
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Started (All patients underwent aggressive resection with intra-operative collection of tissue to generate autologous vaccine. Forty-six patients met all pre- and postoperative criteria for enrollment and constitute the intention-to-treat population) | 70
Completed | 46
Not Completed | 24
Period: Vaccination Treatment Period
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Started | 46
Completed | 46
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Number analyzed (Participants) | 70
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 2
  40-49 years old | 13
  50-59 years old | 19
  60-69 years old | 25
  70-79 years old | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 65
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 70
Median Number of Vaccination Doses Administered [Median (Full Range); unit: vaccine injections] — Population: Only 46 participants were eligible to receive vaccination treatment
  vaccine injections
    number analyzed (Participants) | 46
    (all) | 9 [3 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events of Any Grade
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Number analyzed (Participants) | 46
Participants | 34

2. Primary Outcome: Median Overall Survival
Description: Overall survival is defined as the time from surgical resection to death of any cause.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Number analyzed (Participants) | 46
months | 23.8 [19.8 to 30.2]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the duration of progression-free survival from the time from resection until either documented disease progression or death
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Number analyzed (Participants) | 46
months | 18 [12.4 to 21.8]

4. Secondary Outcome: Median PD-L1 Positivity in Circulating Myeloid Cells
Description: Circulating myeloid cells (CD45+/CD11b+) obtained from patients at the time of surgery were analyzed for PD-L1 expression to determine the percent of myeloid cells positive for PD-L1 (cut off for positivity determined relative to Fluorescence Minus One (FMO) and isotype control).
Time Frame: Up to 53 Weeks
Population: Peripheral blood was available for analysis from 32 vaccine-treated patients
Measure: Median (95% Confidence Interval); unit: percentage of PD-L1 positivity
Arm/Group | Protein Peptide-Complex (HSPPC-96)
Number analyzed (Participants) | 32
percentage of PD-L1 positivity | 54.5 [5.9 to 91.8]

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: Adverse events were reported for the participants who received at least one injection of the vaccine or one dose of temozolomide (TMZ)
Arm/Group | Protein Peptide-Complex (HSPPC-96)
All-Cause Mortality (participants affected / at risk) | 21/46
Serious Adverse Events (participants affected / at risk) | 10/46
Other Adverse Events (participants affected / at risk) | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Protein Peptide-Complex (HSPPC-96) (N=46)
Pain (General disorders) | 1
Seizure (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Protein Peptide-Complex (HSPPC-96) (N=46)
Seizure (Nervous system disorders) | 6 (7)
Ataxia (Nervous system disorders) | 4 (5)
Peripheral motor neuropathy (Nervous system disorders) | 4 (6)
Headache (Nervous system disorders) | 3 (5)
Memory Impairment (Nervous system disorders) | 3 (4)
Nervous system disorders - Other (Nervous system disorders) | 3 (4)
Dysphasia (Nervous system disorders) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Pyramidal tract syndrome (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (28)
White blood cell decreased (Investigations) | 4 (19)
Platelet count decreased (Investigations) | 3 (11)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
CPK increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Fatigue (General disorders) | 6 (14)
Injection site reaction (General disorders) | 16 (16)
Pain (General disorders) | 2 (3)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (3)
Gait disturbance (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (11)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Anemia (Blood and lymphatic system disorders) | 6 (21)
Constipation (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (6)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (4)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes